CLINICAL TRIAL: NCT06458699
Title: Management of Ostomy in Neonates: A Retrospective Single-Center Study
Brief Title: Management Of Stoma In Patients Younger Than 3 Months Old
Acronym: STOMP
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-CF-265
Record Dates: First submitted 2024-06-05; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-04

CONDITIONS: Stoma Colostomy; Stoma Ileostomy; Neonatal Disease
Keywords: Ostomy; Neonate; Outcomes; Costs
MeSH Terms: conditions — Infant, Newborn, Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Hirschsprung's Disease: Patients with Hirschsprung's Disease who had a stoma in the first 3 months of life
- Anorectal MAlformations: Patients with Anorectal MAlformations who had a stoma in the first 3 months of life
- Intestinal Atresia: Patients with Intestinal Atresia who had a stoma in the first 3 months of life
- Necrotizing Enterocolitis: Patients with Necrotizing Enterocolitis who had a stoma in the first 3 months of life
- Intestinal Perforations: Patients with Intestinal Perforations who had a stoma in the first 3 months of life

SUMMARY:
Indications for jejunostomy, ileostomy or colostomy vary in the neonatal population. The most common etiologies are congenital anomalies, such as anorectal malformations, intestinal atresia or Hirschsprung's disease, but also acquired conditions, such as enterocolitis or intestinal perforation. The aim of these stomas is to divert stool in the event of intestinal obstruction or risk of fecal contamination.

Depending on the indication and the type of stoma used, the post-operative follow-up, such as resumption of intestinal transit and feeding, secondary closure of the stoma or not, and the duration and cost of hospitalization differ.

The aim of this study is to compare these differences in order to extract an optimal management strategy, in the light of what is reported in the international scientific literature.

DETAILED DESCRIPTION:
The investigators gathered the data of patients born between January 2009 and December 2023, who had an ostomy made during the first three months of their life.

The investigators then analyzed the patients outcomes ( postoperative complications, length of stay, cost of hospitalization) depending on the etiology of their primary disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had a stoma during the first 3 months of life, from January 2009 to December 2023

Exclusion Criteria:

* Patients who had a stoma after the first 3 months of life, from January 2009 to December 2023
* Patients without a stoma

Ages: 1 Minute to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates whose disease require a stoma during the first 3 months of life, from January 2009 to December 2023
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative medical complications | through study completion, an average of 1 year
  infections, sepsis, dehydration, hydroelectrolytic disorders
Postoperative surgical complications | through study completion, an average of 1 year
  disunion, surgical scar,

SECONDARY OUTCOMES:
Length of stay | through study completion, an average of 1 year
  time of hospitalization
Hospitalization costs | through study completion, an average of 1 year
  costs by department and overall costs

OTHER OUTCOMES:
Redo | through study completion, an average of 1 year
  Necessity to remake the stoma

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Destinval, MD, Study Director — University Hospital, Clermont-Ferrand
Locations (1):
- Clermont-Ferrand University Hospital, Clermont-Ferrand, Auvergne, France